CLINICAL TRIAL: NCT05073302
Title: A Pilot Trial Evaluating a Device-Less Technique in Islet Transplantation
Brief Title: Device-Less Technique in Islet Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00090942
Record Dates: First submitted 2021-02-26; First posted 2021-10-11 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes
Keywords: Device-less, Islet Transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Test a new biomedical intervention in a small group of people for the first time to evaluate safety (e.g. to determine a safe dosage range and to identify side effects)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Implantation of the Device-Less sentinel units. Ultrasound Monitoring. Islet Transplantation. Explantation of Device-Less Sentinels. Standard of Care. Concomitant Care. Post Transplant Testing and Visits. Participant Retention (nine month follow up assessment).
  Interventions: Procedure: Implantation of Nylon catheter (Device-less sentinel unit)

INTERVENTIONS:
Procedure: Implantation of Nylon catheter (Device-less sentinel unit) — Implantation of the Device-Less sentinel units. Ultrasound monitoring will be performed after Device-Less implantation. Standard Islet cell Transplantation: Will occur simultaneously Portal islet transplantation and subcutaneous islet transplantation in the Device-Less sentinel spaces.
  Islets are maintained for a minimum of 6 hours up to 72 hours in supplemented CMRL1066-based media until the time of transplant.
  Concomitant to portal vein infusion, islet transplantation will occur in all four (4) DL sentinel spaces.
  To explant a unit, the Surgeon will make an incision and then carefully dissect the tissue engrafted around the transplant. The entire transplant site and any adherent tissue capsule can then be removed entirely from the pocket.

SUMMARY:
Islet transplantation is an effective modality for treating type 1 diabetes. Despite marked progress in clinical islet transplantation with the achievement and maintenance of insulin independence in over half of recipients up to 5 years, transplant approaches are limited to those that struggle to control their diabetes. Furthermore, this approach remains restricted due to the scarcity of human pancreas donors. While transplanting insulin-producing cells into the liver has been demonstrated as an efficacious means of restoring glycemic control to patients with T1D, the procedure often results in cell loss, and carries risks. Moreover, transplant in to the liver does not permit imaging or retrieval of donor islets. The ability to retrieve the cells is also important for safety reasons.

In theory, the space under the skin is an attractive alternate site for transplanting insulin producing cell, due to ready access, and potential for monitoring cellular transplant function through novel imaging techniques. However, transplantation of insulin producing cells into an unmodified site under the skin universally fails to reverse diabetes in research animal models, or in human studies. Other techniques using devices with different type of technologies and biomaterials have been explored with variable success. Unfortunately, the foreign body and inflammatory reaction persist in the implant. Shapiro Lab, has developed a novel technique called 'device-less' (DL) transplant modality. This approach was designed to harness an innate foreign body response in a favorable and controlled manner, to induce growth of new blood vessels to allow the survival of the insulin producing cells without the natural body response to foreign body. Briefly, this site transforms the inhospitable under the skin site into a viable location through the temporary implantation of a small tube called angiocatheter.

For this study, 5 patients will received transplant in to the modified site under the skin using the DL transplant technique.

DETAILED DESCRIPTION:
1. Before any study-specific procedure is performed, valid informed consent will be obtained.
2. A complete medical history will be collected including smoking status and alcohol frequency.

   On admission to hospital, the recipient will be assessed for fitness to proceed to transplant according to local procedures. If a recipient is deemed unfit for transplant at the time of admission, they will no longer be active on the transplant waiting list and as such will be excluded from the trial.
3. Implantation of the DL sentinel unit: Occurs at Visit 3 (2 Weeks to 24 Weeks Prior to Islet Transplant). One DL sentinel unit will be implanted in the forearm, as deemed appropriate by the Investigator. To conduct the procedure, local anesthesia with sedation may be utilized, with use of general anesthesia at the discretion of the Surgeon. Implantation is executed via incision followed by formation of tissue pockets for each DL unit. Incisions are up to approximately 10 to 30 mm in length, but could vary. The DL unit will consist of a minimum of 5 French (Fr) or up to 7 Fr Torcon NB® Advantage nylon catheters prepared to 8-10 cm in length. Each DL unit will be inserted into one subcutaneous pocket prepared. Surgeons trained on the procedure will have discretion on the ultimate number and length of incisions, but should discuss the details of the implantation plan with the subject prior to the surgery.

   * There are inherent surgical risks with the implantation and explantation of DL sentinel units including pain, bleeding, hematoma, seroma, tenderness, redness, scarring, and infection. Steps will be taken to minimize the risks and to make the subject comfortable during the procedure with anesthetic and post-procedure analgesia.
   * With any implanted product, the possibility of migration or extrusion of the DL implant exists.
   * The use of anesthesia itself may cause side effects. The type(s) of anesthesia used during the implantation and explantation procedures will be determined by the Investigator. Side effects may include, but are not limited to:

     * Local Anesthesia: Stinging and/or a burning sensation. Less likely side effects include nausea, vomiting, dizziness, drowsiness, allergic reactions (e.g., redness, itching, and rash), low blood pressure, weakness, severe numbness or tingling, ringing in ears, blurry or double vision, slurred speech, metallic taste in the mouth, mental status change, muscle twitching, and seizures.
     * General Anesthesia: Harm to the vocal cords, heart attack, lung infection, and stroke, trauma to the teeth or tongue, or temporary mental confusion. Rarely, waking during anesthesia or death may occur.
     * Conscious Sedation: Difficulty breathing.
4. Ultrasound Monitoring Ultrasound monitoring will be performed after DL implantation as per the Principal Investigator's discretion.
5. Standard Islet cell Transplantation: Will occur simultaneously Portal islet transplantation and subcutaneous islet transplantation in the DL sentinel spaces.

   Standard islet isolation procedures will be followed for all aspects of the islet isolation process. The final islet product will be evaluated based on standard assays used in standard islet isolation practice. Islet transplantation occurs at Visit 4 (Day 0).

   A minimum target of 4,000 IEQ/kg recipient body weight will be infused either via a percutaneous transhepatic catheter inserted into the portal vein under ultrasound and fluoroscopic guidance, or by open laparotomy under general anesthesia (via cannulation of an omental or mesenteric vein), at the discretion of the investigators. Islets are maintained for a minimum of 6 hours up to 72 hours in supplemented CMRL1066-based media until the time of transplant. The packed islet tissue volume preparation will not exceed 10 cc in order to minimize the risk of portal thrombosis and post-procedural bleeding. Islet transplant into the portal vein is part of Alberta Health Services standard of care procedures.

   Concomitant to portal vein infusion, islet transplantation will occur in the DL sentinel space. A small incision will be made cranial to the implanted DL unit. A small section of implanted catheter is cut to expose the vascularized tissue scaffold. The DL unit is exposed through the superficial incision and PE-50 or PE-90 tubing containing the human islet preparation is inserted into the lumen of the DL catheter. Approximately 500 - 4000 Islet Equivalent (IEQ), equivalent to 20 μl of islet tissue, will be infused into the DL sentinel. This is based on the original islet mass and packed tissue volume before transplantation and the volume of 8 cm of PE-50 tubing with 0.53 mm inner diameter. The DL catheter is subsequently withdrawn along the PE-50 (or PE-90) tubing and the islets are subsequently infused into the resulting DL lumen.
6. Explantation of DL Sentinels: One quarter of the DL sentinel will be explanted at 2, 4, 12, and 24 weeks post islet transplant, respectively. Experiences in other studies investigating subcutaneous transplantation indicate that while under anesthesia, the units and the surrounding tissue can be explanted with traditional surgical instruments. Local anesthesia is required at a minimum, with the use of sedation or general anesthesia at the discretion of the Surgeon. To explant a unit, the Surgeon will make an incision (re-entry thru the same implant/transplant incision is advocated) and then carefully dissect the tissue engrafted around the transplant. The entire transplant site and any adherent tissue capsule can then be removed entirely from the pocket.

As this is a first in human study, there is the possibility the explantation procedure and technique will be modified based on the data collected.

Participants may receive all required concomitant medications for islet transplant patients: Alemtuzumab, basiliximab, tacrolimus, mycophenolate mofetil, etanercept and anakinra are Standard of Care medications used in the Clinical Islet Transplant program.

Participants in the study receiving their islet transplants will be managed following standard of care including implantation procedure, peri- and post-operative care, post-transplant monitoring, immunosuppression and other medications. For detailed islet transplant standard of care (pre- and post- islet transplant assessments and evaluations), please refer to Appendix B of the study protocol.

7. Portions of the same device-less (DL) biopsy samples will be assessed by histology and MMDx approaches. MMDx assessments of explanted tissue are standardized molecular measurements (probabilities) of transplant rejection or injury.

No additional samples will be required. Samples sent to the (ATAGC) will be coded by the trial personnel. The only required information will be the time of DL explant, post implantation. There will be no additional risks for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Reduced awareness of hypoglycemia, as defined by the absence of adequate autonomic symptoms at plasma glucose levels < 3.0 mmol/L, indicated by, 1 or more episodes of severe hypoglycemia requiring third-party assistance within 12 months, a Clarke score ≥4, HYPO score ≥1,000, lability index (LI) ≥400 or combined HYPO/LI >400/>300.
* Metabolic instability, characterized by erratic blood glucose levels that interfere with daily activities and/or 1 or more hospital visits for diabetic ketoacidosis over the last 12 months.
* Participants must be capable of understanding the purpose and risks of the study and must sign a statement of informed consent.

Exclusion Criteria:

* Significant skin conditions involving the area(s) targeted for implantation. Examples include but are not limited to recurrent boils/furuncles, extensive surgery or scarring, or lipodystrophy.
* History of enrollment in any other islet transplant trials and islet transplant under standard of care (at the discretion of the investigator).
* Severe co-existing cardiac disease, characterized by any one of these conditions: (a) recent (within the past 6months) myocardial infarction; (b) left ventricular ejection fraction <30%; or (c) evidence of ischemia on functional cardiac exam.
* Active alcohol or substance abuse, including cigarette smoking (must be abstinent for 6 months prior to listing for transplant).
* Psychiatric disorder making the subject not a suitable candidate for transplantation (e.g., schizophrenia, bipolar disorder, or major depression that is unstable or uncontrolled on current medication).
* History of non-adherence to prescribed regimens.
* Active infection including Hepatitis C, Hepatitis B, HIV, or TB (subjects with a positive PPD performed within one year of enrollment, and no history of adequate chemoprophylaxis).
* Any history of, or current malignancies except squamous or basal skin cancer.
* BMI > 35 kg/m2 at screening visit.
* Age less than 18 or greater than 68 years.
* Measured glomerular filtration rate (GFR) <60 mL/min/1.73 m2.
* Presence or history of macroalbuminuria (>300 mg/g creatinine).
* Clinical suspicion of nephritic (hematuria, active urinary sediment) or rapidly progressing renal impairment (e.g. Increase in serum creatinine of 25% within the last 3-6 months).
* Baseline Hb < 105 g/L (<10.5 g/dL) in women, or < 120 g/L (<12 g/dL) in men.
* Baseline screening liver function tests outside of normal range, with the exception of uncomplicated Gilbert's Syndrome. An initial LFT panel with any values >1.5 times the upper limit of normal (ULN) will exclude a patient without a re-test; a re-test for any values between ULN and 1.5 times ULN should be made, and if the values remain elevated above normal limits, the patient will be excluded.
* Untreated proliferative retinopathy.
* Positive pregnancy test, intent for future pregnancy or male subjects' intent to procreate, failure to follow effective contraceptive measures, or presently breast-feeding.
* Evidence of significant sensitization on PRA (at the discretion of the investigator).
* Insulin requirement >1.0 U/kg/day
* HbA1C >12%.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Rate of Adverse Events/Serious Adverse Events | 9 months
  Adverse Events/ Serious Adverse Event experienced by the participants in the study
Rate of inflammation in the DL implant site | 9 months
  Implant tolerability assessment

SECONDARY OUTCOMES:
Probability of rejection or injury analyzed using the Molecular Microscope Diagnostic System (MMDx) system by measuring the expressions of all genes within the graft | 9 months
  Molecular Microscope Diagnostic System (MMDx) of the explanted tissue
Percentage of live cells measured by immunohistochemistry | 9 months
Presence of vascularization demonstrated by immunohistochemistry | 9 months
Presence of immune response demonstrated by immunohistochemistry | 9 months
Cellular composition demonstrated by immunohistochemistry | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: James Shapiro, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Clinical Islet Transplant Program, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: related link — http://www.islet.ca/